CLINICAL TRIAL: NCT03592797
Title: Effect of Laser Acupuncture Treatment on Chronic Facial Paralysis: A Randomized Sham Control, Double Blind Pilot Study
Brief Title: Effect of Laser Acupuncture Treatment on Chronic Facial Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH107-REC1-030
Record Dates: First submitted 2018-06-11; First posted 2018-07-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Bell Palsy; Idiopathic Facial Paralyses
Keywords: Low-level laser therapy; Laser acupuncture; Sequelae of Bell's palsy; Randomized controlled trial
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Intervention Model Description: Randomized, sham control, double blind pilot study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham laser acupuncture group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser acupuncture therapy group (Experimental): Each subject in the experimental group will receive laser acupuncture therapy using Handylaser Trion device (RJ Laser, Germany) to stimulate acupuncture points with laser beam irradiation.
  Interventions: Other: Laser acupuncture therapy
- Sham laser acupuncture therapy group (Sham Comparator): Each subject in the sham control group will receive laser acupuncture therapy using Handylaser Trion device (RJ Laser, Germany). The laser device in the sham group will be deactivated and won't produce any laser beam irradiation on acupuncture points
  Interventions: Other: Sham laser acupuncture therapy

INTERVENTIONS:
Other: Laser acupuncture therapy — Low level laser therapy to stimulate acupuncture points: Total 11 points will be used in the study. 7 points ST4, ST6, ST7, SI18, BL2, GB14, SJ17 located in the effected side of the face and will be stimulated ipsilateral. Two points ST36, LI4 located distally and will be stimulated bilateral.
  Arms: Laser acupuncture therapy group
Other: Sham laser acupuncture therapy — Sham procedure of Low level laser therapy to stimulate acupuncture points is identical procedure as the intervention group. The same 11 points which mention above will be used, However, in the sham group the laser device will be deactivated and won't produce any laser beam irradiation.
  Arms: Sham laser acupuncture therapy group

SUMMARY:
Inadequate recovery from Bell's palsy is not uncommon and as consequence, physical and social impairment are exist in these patients. The medical options for chronic condition of Bell's palsy are insufficient. Low-level laser therapy has shown a favorable prognosis in the regeneration of peripheral nerves. Moreover, laser acupuncture therapy (LAT) become widely used method to stimulate acupuncture points, but its efficacy as treatment method for Bell's palsy and during the chronic stage is unclear.

DETAILED DESCRIPTION:
Background: Inadequate recovery from Bell's palsy is not uncommon and as consequence, physical and social impairment are exist in these patients. The medical options for chronic condition of Bell's palsy are insufficient. Low-level laser therapy has shown a favorable prognosis in the regeneration of peripheral nerves. Moreover, laser acupuncture therapy (LAT) become widely used method to stimulate acupuncture points, but its efficacy as treatment method for Bell's palsy and during the chronic stage is unclear.

Methods: This clinical trial settings are a randomized, placebo control, double blind pilot study including patients with the unsatisfactory recovery of Bell's palsy with the following two groups: LAT (N=16) and a sham LAT (N=16). The LAT will receive treatments for 6 weeks, compare to sham control group. The primary outcome measure will be change in the Facial Disability Index at week 6. Statistical analysis will also include changes in the House-Brackmann grading system, the Sunnybrook grading system and stiffness scale at 1, 3 and 6 weeks after randomization.

Expected outcome: The investigators hypothesis that LAT will have an effect on functional outcomes in patients with chronic facial paralysis. Moreover, changes in the S-B facial nerve grading system is also expected to have an improvement. Last, social subscale of FDI is expected to have an improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed patients with Bell's palsy (ICD9- CM 351.0) with at least 3 months prior to screening.
2. Age- above 20 years old
3. Facial disability index (FDI) less than 80 on FDI physical subscale and less than 80 on the FDI social subscale.

Exclusion Criteria:

1. Patients with any of the following are excluded: uncontrolled hypertension, diabetes mellitus requiring insulin injection, other neurological diseases, patients with multiple cranial nerve palsies, pregnancy or breastfeeding woman, will be excluded.
2. Patients with other types of facial palsy or other known causes than Bell's palsy-Ramsay Hunt syndrome, cholesteatoma, Otitis media, traumatic facial palsy, iatrogenic facial palsy or parotid tumor will be excluded.
3. Patients with recurrent facial palsy or patients who have pre-existing facial deformity, contracture, synkinesis, and spasm for whatever reason will be excluded.
4. Patients with the following will be excluded:

Surgery: a surgical history for facial palsy, such as facial nerve decompression, reconstruction of the facial nerve or muscle within 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
The change in the Facial Disability Index (FDI) | Assessment will take place at baseline, end of third week and six week.
  The primary outcome measurement in this study is the change of FDI after completing 6 weeks of laser acupuncture therapy. FDI scoring system consists of two domains; physical score and social score and each section consists five multiple choice question related to either physical or social issues occurred in the previous month. Subjects will fill up the questionnaire and the assessor will calculate the score according to the calculation in each section; physical section: total score (questions 1--5) minus N divided by N multiple 100 divided 4 equals to total score. social section; total score (questions 6--10) minus N divided by N multiple 100 divided by 5 equals to total score (N equals to number of questions answered). Higher values represent a better outcome. FDI evaluations will be performed on the first visit, the 9th visit and 18th visit and will be compared to the score at baseline.

SECONDARY OUTCOMES:
The change in the House-Brackmann (H-B) facial nerve grading system | Assessment will take place at baseline, end of third week and six week.
  The change of H-B facial nerve grading system will be compared after completing 6 weeks of laser acupuncture therapy. H-B facial nerve grading system includes 6 grades of facial paralysis; normal, mild, moderate, moderate severe, severe and complete paralysis. The study assessor asks the patient to move the facial muscles and then according to the result the assessor decides the grade of paralysis. The evaluations will be performed on the first visit, the 9th visit and 18th visit.
The change in the Sunnybrook (S-B) facial nerve grading system | Assessment will take place at baseline, end of third week and six week.
  The change of S-B facial nerve grading system will be compared after completing 6 weeks of laser acupuncture therapy. S-B facial nerve grading system includes 3 subscales; resting symmetry (eye, cheek and mouth), symmetry of voluntary muscles and synkinesis. Besides the resting symmetry, in the two others subscales the assessor asks the patient to move the facial muscles and then give a score between 1 to 5 ( 1= unable to move 5= complete moment). Subscales are combined to compute a total score; symmetry of voluntary muscles subscale minus resting symmetry subscale minus synkinesis subscale equals to total score. Higher values represent a better outcome. The evaluations will be performed on the first visit, the 9th visit and 18th visit.
The change in the stiffness scale | Assessment will take place at baseline and end of six week.
  The change of the stiffness score will be compared to baseline. The stiffness scale will be hand in each session and the subject will choose one number from a five-point scale (1= no stiffness to 5= very stiff) according to the feeling in the face after receiving laser acupuncture therapy. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, M.D PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ton G, Lee LW, Ng HP, Liao HY, Chen YH, Tu CH, Tseng CH, Ho WC, Lee YC. Efficacy of laser acupuncture for patients with chronic Bell's palsy: A study protocol for a randomized, double-blind, sham-controlled pilot trial. Medicine (Baltimore). 2019 Apr;98(15):e15120. doi: 10.1097/MD.0000000000015120. PMID 30985671